CLINICAL TRIAL: NCT03388827
Title: The Use of Laminaria Versus Laminaria Plus Misoprostol Before Operative Hysteroscopy in Nulliparous Women . A Double Blinded Randomized Trial.
Brief Title: Laminaria and Misoprostol Before Operative Hysteroscopy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, IBRAHIM ABD ELGAFOR, assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZUH- 9
Record Dates: First submitted 2017-12-25; First posted 2018-01-03 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2017-12

CONDITIONS: Cervical Spasm
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laminaria (Experimental): Laminaria tent was introduced in the cervical canal
  Interventions: Device: Laminaria tent
- Laminaria plus Misoprostol (Active Comparator): Laminaria and Misoprostol were introduced
  Interventions: Drug: Laminaria plus Misoprostol

INTERVENTIONS:
Device: Laminaria tent — Laminaria tent was inserted for 12 hours before Hysteroscopy
  Arms: Laminaria
Drug: Laminaria plus Misoprostol — Laminaria plus Misoprostol were inserted for 12 hours before Hysteroscopy
  Other Names: cytotec,
  Arms: Laminaria plus Misoprostol

SUMMARY:
Laminaria and Misoprostol before Operative Hysteroscopy

DETAILED DESCRIPTION:
The use of laminaria versus laminaria plus misoprostol was compared before operative hysteroscopy in nulliparous women to assess the efficacy of both methods in cervical dilatation.

ELIGIBILITY:
Inclusion Criteria: nullipara

* need hystroscopic intervention

Exclusion Criteria: previous pregnancy

cervical lesion

contraindication to misoprostol

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Preoperative cervical width | 12 hours
  cervical width in Hegar dilators number

SECONDARY OUTCOMES:
adverse effects | 24 hours
  adverse effects of the method used or hysteroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided